CLINICAL TRIAL: NCT02680171
Title: Feasibility and Effectiveness Study of Implementing Prism Adaptation as a Treatment for Spatial Neglect After Right Hemisphere Stroke
Brief Title: Feasibility and Effectiveness Study of Implementing Prism Adaptation as a Treatment for Spatial Neglect After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Gail Eskes, Dr., Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRICSpatialNeglect2016
Record Dates: First submitted 2016-01-27; First posted 2016-02-11 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Sensory Neglect; Stroke
Keywords: Cognitive Rehabilitation; Prism Adaptation; Stroke; Spatial Neglect
MeSH Terms: conditions — Perceptual Disorders; Stroke

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prism adaptation treatment (Experimental): Prism Goggles with ten-degree rightward deviating prism lenses will be used to implement prism adaptation treatment, in addition to standard care.
  Interventions: Behavioral: Prism Goggles
- Sham prism adaptation treatment (Sham Comparator): Non-Shifting Goggles (sham) will be worn by patients in the control condition. These goggles do not shift the patients visual field.
  Interventions: Other: Non-Shifting Goggles

INTERVENTIONS:
Behavioral: Prism Goggles — Patients in the experimental condition will wear prism goggles while completing a computerized aiming task. This prisms will shift the patients' vision 10 degrees rightward, causing a recalibration of visuo-motor information. Prism adaptation will be carried out over several days.
  Arms: Prism adaptation treatment
Other: Non-Shifting Goggles — Non-shifting goggles are worn instead of prism goggles, while completing the same computerized aiming task as those assigned to the prism adaptation.
  Other Names: Control condition
  Arms: Sham prism adaptation treatment

SUMMARY:
Spatial neglect is a common attention disorder after right hemisphere stroke and is associated with decreased independence and quality of life. Despite its high prevalence in the stroke population, there is currently no standard of care for the treatment of neglect. Prism adaptation (PA) is a promising rehabilitation technique, however incorporation into clinical care has been limited likely due to the lack of standardized procedures. The investigators have developed a computerized PA technique designed to better engage patients and assist clinicians. In this study the investigators aim to evaluate the feasibility and effectiveness of the computerized PA procedure in a typical health care setting, with the hypothesis that the PA procedure will improve patient's neglect symptoms.

DETAILED DESCRIPTION:
There is an unmet need for effective and feasible interventions for spatial neglect after right hemisphere stroke. Neglect is a frequent problem after stroke and makes it difficult for individuals to pay attention and notice information coming from the left side of their world. Thus, they often miss food on the left side of their plate, fail to wash or groom the left side of their face or body, or run into objects on the left side of the hall when walking or using their wheelchair. Neglect is associated with slower recovery, reduced independence, longer stays in rehabilitation and need for more resources when discharged. The investigators have developed a novel and simple computerized prism adaptation (PA) procedure for treating neglect, but the investigators don't know yet whether it is feasible and effective in a typical health care setting. Thus, the purpose of this project is to conduct a randomized, controlled clinical trial, comparing the PA method to a control intervention for the treatment of neglect. The investigators will measure feasibility of use in a clinical setting and effectiveness in terms of impairment (i.e., does PA improve neglect symptoms?), activities (i.e., does having PA improve independence in daily activities) and health care outcomes (i.e., does giving PA shorten length of stay and decrease the need for resources on discharge?). By treating neglect with PA, the overall aim is to improve the health care outcomes for those with neglect and to reduce need for extended hospital care.

A controlled, randomized design will be used in the present study. Patients will be randomly assigned (with stratification related to neglect severity) to PA (experimental) or sham (control) conditions and complete 10, 30-minute intervention sessions over approximately two weeks. These intervention sessions will involve a novel and simple computerized prism adaptation, Peg-The-Mole (PTM). Outcome measures will be collected before and after each treatment, as well as at baseline, and a three month follow-up over the phone.

ELIGIBILITY:
Inclusion Criteria:

* Experience mild to severe symptoms of neglect (as measured by the Sunnybrook Neglect Assessment Procedure and/or as determined based on clinical judgment of the treating team)
* Be willing to participate
* Be able to consent to participate
* Be medically stable
* Have normal or corrected to normal vision
* Be able to point to targets presented on a computer screen.

Exclusion Criteria:

* Other neurological disease (e.g., Multiple Sclerosis, Parkinsons disease)
* Dementia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Sunnybrook Neglect Assessment Procedure (SNAP) | Taken at baseline and after the intervention has been completed (approximately two weeks post-treatment start)
  Test of neglect severity

SECONDARY OUTCOMES:
Change in Johnny Shirt Visual Scanning Task | Taken at baseline, after five intervention sessions are completed (approximately 1 week post-treatment start), and after the intervention (approximately two weeks post-treatment start)
  Test of neglect severity
Change in Behavioural Inattention Test - Behaviour subtests (BIT-B) | Taken at baseline and after the intervention (approximately two weeks post-treatment start)
  Test of neglect severity
Change in Catherine Bergego Scale (CBS) | Taken at baseline and after the intervention (approximately two weeks post-treatment start)
  Scale of neglect impact on daily activities
Change in Halifax Neglect Severity Scale | Taken after the intervention (approximately two weeks post-treatment start) and at follow-up (approximately 3 months post-discharge from the Nova Scotia Rehabilitation and Arthritis Centre)
  Scale of neglect impact on daily activities
Change in Functional Independence Measure (FIM) | Taken at baseline and at discharge up to 3 months
  Measure of functional independence
Frenchay Activities Index | Taken at approximately 3 months post-discharge
  Measure of functional independence
Length of inpatient stay at the Rehabilitation Centre | From admission to discharge up to 3 months
  Measure of hospital utilization
Discharge destination from Rehabilitation Centre | At time of discharge up to 3 months from admission
  Measure of hospital utilization
Change in Proprioceptive and Visuo-motor pointing midline tasks | Taken from immediately before and at end of treatment session, about 10 minutes
  Used to assess prism adaptation after-effects

CONTACTS AND LOCATIONS:
Overall Officials: Gail A Eskes, PhD, Principal Investigator — Nova Scotia Health Authority; Dalhousie University; Richard Braha, PhD, Principal Investigator — Nova Scotia Health Authority; Anne Sophie Champod, PhD, Study Chair — Dalhousie University; Acadia University; Joy Boyce, BScOT, Study Chair — Nova Scotia Health Authority; Myrna King, BScOT, Study Chair — Nova Scotia Health Authority
Locations (1):
- Nova Scotia Health Authority, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Champod AS, Taylor K, Eskes GA. Development of a new computerized prism adaptation procedure for visuo-spatial neglect. J Neurosci Methods. 2014 Sep 30;235:65-75. doi: 10.1016/j.jneumeth.2014.05.023. Epub 2014 Jun 19. PMID 24952321
- [Derived] Longley V, Hazelton C, Heal C, Pollock A, Woodward-Nutt K, Mitchell C, Pobric G, Vail A, Bowen A. Non-pharmacological interventions for spatial neglect or inattention following stroke and other non-progressive brain injury. Cochrane Database Syst Rev. 2021 Jul 1;7(7):CD003586. doi: 10.1002/14651858.CD003586.pub4. PMID 34196963